CLINICAL TRIAL: NCT03136575
Title: The Impact of the Digital Traditional Qigong Regimen Exercises on Quality of Life and Sleep Disturbance in Head and Neck Patients Undergoing Radiotherapy
Brief Title: The Impact of Qigong on Quality of Life and Sleep Disturbance in Head and Neck Patients Undergoing Radiotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Collaborators: Kaohsiung Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KMUHIRB-E(II)20150219
Record Dates: First submitted 2017-04-20; First posted 2017-05-02 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Qigong

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant
Masking Description: patients who signed inform consent are randomized into qigong group and wait-list control (WLC)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Qigong (Active Comparator): Patients in the Qigong group receive Qigong,a mind-body exercise, 3 times a week, for 6 weeks during radiotherapy course. The participants are given a DVD contains Qigong program, and they attend the Qigong class in a health education room at the radiation oncology department to assure their attendance.
  Interventions: Behavioral: Qigong
- wait-list control (Placebo Comparator): Patients who are assigned to the wait-list control are told to have some exercise by their own but no actually attend the the class in fact.
  Interventions: Behavioral: Wait-list control

INTERVENTIONS:
Behavioral: Qigong — a 30 minutes exercise program, 3 times a week and lasts for 6 weeks during radiotherapy course
  Arms: Qigong
Behavioral: Wait-list control — patients enrolled in this group are informed orally to have exercise only and are arranged in a waiting list
  Arms: wait-list control

SUMMARY:
This study aimed to observe how a six week qigong program influence patients with head and neck cancer during active radiotherapy treatment course. The quality of life, sleep dysfunction or depression and shoulder and neck function will be accessed by questionnaire, and ANS function will be objectively investigated using heart rate variability measurement.

DETAILED DESCRIPTION:
The incidence of head and neck cancers is the 6th in Taiwan, and head and neck cancers are the 5th leading cause of cancer death, causing approximately 2000 death in 2010. Head and neck cancers patients usually require multimodality treatments, including surgery, chemotherapy and radiotherapy. These treatments can cause functional deterioration and worsened quality of life during or after the treatment, and bring tremendous effects on patient's life. When radiotherapy is indicated, it requires 6 to 7 weeks treatment, and most patients suffered from different degrees of mucositis, dermatitis, xerostomia and neck and shoulder tightness during radiotherapy. How to improve quality of life for these patients during radiotherapy is an important task.

Qigong is a mind-body exercise or therapy; it can improve quality of life, such as fatigue, sleep dysfunction and depression through regulation of breath and simple physical exercise. Some found that the qigong can decrease inflammation and show some impact on accommodation of ANS in cancer patients. Most studies focus on how qigong effect on cancer survivors, however, this study is aimed to observe how a six week qigong program influence patients with head and neck cancer during active radiotherapy treatment course. The quality of life, sleep dysfunction or depression and shoulder and neck function will be accessed by questionnaire, and ANS function will be objectively investigated using heart rate variability measurement.

ELIGIBILITY:
Inclusion Criteria:

- Clinical diagnosis of Head and neck squamous cell carcinoma, subsites including nasopharyngeal cancer, oropharyngeal cancer, oral cancer, hypopharyngeal cancer and laryngeal cancer Performance status ECOG 0-1 Physically able to participate in the qigong program

Exclusion Criteria:

- Previous radiotherapy to head and neck region Patients who refused to sign the informed consents Patients who took antihypertensive drugs, sedatives, or antiarrhythmic drugs

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 90% of head and neck cancer patients are male gender, so this study mainly includes male
Enrollment: 60 (Estimated)
Dates: Start 2016-03-28 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of quality of life | before radiotherapy starts and after radiotherapy complete. (The duration of radiotherapy course is usually about 6 to 7 weeks)
  The changes of quality of life before radiotherapy and after radiotherapy complete are evaluated using University of Washington Quality of Life Questionnaire (UW-QOL) to access the quality of life
Change of depression and anxiety | before radiotherapy start and after radiotherapy complete. (The duration of radiotherapy course is usually about 6 to 7 weeks)
  The changes of the level of depression and anxiety before radiotherapy and after radiotherapy complete are accessed using hospital anxiety and depression scale (HADS)
Change of sleep quality | before radiotherapy start and after radiotherapy complete (The duration of radiotherapy course is usually about 6 to 7 weeks)
  The change of sleep quality is evaluated using Pittsburgh Sleep Quality Index (PSQI)
Change of Autonomic nervous system (ANS) function | before radiotherapy start and after radiotherapy complete(The duration of radiotherapy course is usually about 6 to 7 weeks)
  The change of ANS function is accessed by heart rate variability

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsihung Medical University Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No